CLINICAL TRIAL: NCT05041296
Title: The Epileptic Heart - Multiparametric Cardiac Magnetic Resonance Imaging for Detection and Quantification of Acute and Chronic Cardiac Involvement in Patients With Epilepsy
Brief Title: Cardiac MRI for Detection of Acute and Chronic Cardiac Involvement in Patients With Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Julian Alexander Luetkens, Principal Investigator, Senior Physician, University Hospital, Bonn
Other Study IDs: 534/20
Record Dates: First submitted 2021-08-27; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Epilepsy; Cardiomyopathies
MeSH Terms: conditions — Epilepsy; Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic group: Chronic epilepsy with recurrent seizures
  Interventions: Diagnostic Test: Cardiac magnetic resonance scan
- Acute group: Epilepsy and short-term history of seizures
  Interventions: Diagnostic Test: Cardiac magnetic resonance scan
- Control group: Healthy participants
  Interventions: Diagnostic Test: Cardiac magnetic resonance scan

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance scan — Multiparametric cardiac magnetic resonance including traditional and quantitative functional and structural parameters

SUMMARY:
The aim of the study is to use multiparametric cardiac MRI to identify any abnormalities in myocardial structure and function in patients with epilepsy. A two-stage study design is planned as part of the study:

1. In the acute setting, cardiac MRI will be performed in patients before and after a tonic-clonic seizure and compared intraindividually. In this study arm, potential acute seizure-induced myocardial damage will be detected.
2. In the chronic setting, cardiac MRI will be performed in patients with known chronic epilepsy during the seizure-free interval to detect potential chronic myocardial damage (myocardial fibrosis) and compared with a control population. Within the group of epilepsy patients, possible associations with various epilepsy-specific characteristics (e.g., form, cause, onset, duration, and severity of epilepsy) will be investigated.

ELIGIBILITY:
Inclusion criteria:

1. diagnosed epilepsy
2. examination under usual antiepileptic pharmacotherapy or medication up-dosing (if medication was reduced during video-EEG recording)
3. age between 18-60 years

Exclusion criteria:

1. underlying cardiac disease, e.g. coronary artery disease, previous myocardial infarction, previous myocarditis, complex congenital heart defect, known cardiomyopathy of other cause
2. pregnant and breastfeeding women
3. patients who use IUD for contraception
4. patients with a contraindication to contrast enhanced MRI

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients with epilepsy with treatment in the Clinic and Polyclinic for Epileptology of the University Hospital Bonn (Primary care clinic)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
T1 relaxation time | Measurement will be performed within 2 weeks after MRI scan.
  T1 relaxation times will be obtained to asses acute myocardial injury and fibrosis. T1 maps will be analyzed using a segmental approach by region of interest analysis. T1 relaxation times are given in [ms].

SECONDARY OUTCOMES:
T2 relaxation time | Measurement will be performed within 2 weeks after MRI scan.
  T2 relaxation times will be obtained to asses myocardial edema. T2 maps will be analyzed using a segmental approach by region of interest analysis. T2 relaxation times are given in [ms].
Extracellular volume fraction | Measurement will be performed within 2 weeks after MRI scan.
  Myocardial extracellular volume will be obtained to asses extracellular space/myocardial fibrosis. ECV values will be calculated using a segmental approach by region of interest analysis of native and contrast-enhanced T1 relaxation maps. ECV values are given in [%].
Myocardial strain | Measurement will be performed within 2 weeks after MRI scan.
  Cardiac magnetic resonance feature-tracking will be used to asses left ventricular longitudinal, circumferential and radial strain (Strain values are given in [%]).

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Bonn, Clinic and Polyclinic for Epileptology, Bonn, North Rhine-Westphalia
  - University Hospital Bonn, Clinic for Diagnostic and Interventional Radiology, Bonn, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No